CLINICAL TRIAL: NCT05700708
Title: Point-of-Care Echocardiography to Assess Impact of Dynamic Cardiac Function, Renal and Cardiac Biomarkers in Cirrhosis With Refractory Ascites
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: NK-2020-2141
Record Dates: First submitted 2022-12-06; First posted 2023-01-26 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Cirrhosis, Liver; Acute-On-Chronic Liver Failure; Refractory Ascites; Ascites; Acute Kidney Injury
Keywords: Ascites; Cirrhotic Cardiomyopathy; Acute kidney injury
MeSH Terms: conditions — Liver Cirrhosis; Acute-On-Chronic Liver Failure; Ascites; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cirrhosis with Refractory Ascites
  Interventions: Diagnostic Test: Echocardiographic assessment

INTERVENTIONS:
Diagnostic Test: Echocardiographic assessment — POC-Echocardiography to assess dynamic changes in cardiac output to assess therapeutic responses with albumin, midodrine, diuretics and domiciliary albumin

SUMMARY:
Point-of-care echocardiography (POC-Echo) is used to determine left ventricular systolic and diastolic dysfunction (LVDD), inferior vena cava (IVC) dynamics and volume status in cirrhosis and Acute-on-chronic liver failure ACLF accurately.

We will assess IVC dynamics, LV systolic function [LV ejection fraction (EF) & cardiac output (CO)], and diastolic dysfunction (E/e', e' and E/A ratio) and urinary biomarkers (cystatin C and NGAL) in patients with cirrhosis and Refractory Ascites.

DETAILED DESCRIPTION:
The decrease in systemic vascular resistance (SVR) and redistribution of blood volume with reduced intravascular volume compartment and third space fluid losses. Systemic vasodilatation is compensated by an increase in cardiac output (CO) in the initial stages of compensated cirrhosis. However, as the stage of liver cirrhosis progresses to decompensation, more prominent arterial vasodilatation and reduced SVR leads to a fall in CO. Thus, the cardiac homeostat is reset in a cirrhotic hyperdynamic circulation, wherein an increased heart rate, and therefore, increased cardiac output will no longer be able to compensate for the reduced mean arterial pressure (MAP), and decreased blood volumes in central venous territories.18 Consequent activation of vasoconstrictor systems including renin-angiotensin-aldosterone, vasopressin and the sympathetic nervous system comes into play to maintain the intravascular blood volume and pressure. These compensatory pathways cause an increase in sodium and water retention resulting in refractory ascites and hepatorenal syndrome (HRS). In critically ill patients with cirrhosis, the limited cardiac reserve is further stressed, CCM and heart failure may be diagnosed for the first time when the patient develops sepsis or septic shock.

Point-of-care echocardiography (POC-Echo) is used to determine left ventricular systolic and diastolic dysfunction (LVDD), inferior vena cava (IVC) dynamics and volume status in cirrhosis accurately. We will assess IVC dynamics, LV systolic function [LV ejection fraction (EF) & cardiac output (CO)], and diastolic dysfunction (E/e', e' and E/A ratio) in patients with cirrhosis ACLF and refractory ascites

Definition of CCM is as per updated CCMC criteria of 2020.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis of any Etiology
* Patient with Refractory Ascites

Exclusion Criteria:

* Hepatocellular carcinoma
* Patients with active variceal bleeding
* HIV or severe immunocompromised state
* Chronic kidney disease (CKD) on renal replacement therapy (RRT),
* Previous transjugular intra hepatic portosystemic shunt (TIPS)
* Porto-pulmonary hypertension,
* Coronary artery disease
* Congenital or valvular heart disease
* Prosthetic cardiac valves

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhosis of any etiology, aged between 18-65 years, with Refractory Ascites definition as per International Ascites club.
  1. Diuretic-resistant ascites
  2. Diuretic-intractable ascites
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Cardiac output measurement by echocardiography after albumin | Day 0
  Echocardiographic assessment of cardiac output in L/min will be recorded at least 3 time points, day 0, day 1 and day 2.
  The cardiac output at 3 days after enrollment and albumin therapy will also be documented. The Doppler velocity time integral (VTI) method in estimating stroke volume and cardiac output correlates well with results of concurrent thermodilution cardiac output determinations in patients without significant left-sided valvular regurgitation.
  Cardiac output(CO), Stroke volume (SV), Heart rate (HR)
  CO = [SV * HR]/ 1000
Cardiac output measurement by echocardiography after albumin | Day 1
  Echocardiographic assessment of cardiac output in L/min will be recorded at least 3 time points, day 0, day 1 and day 2.
  The cardiac output at 3 days after enrollment and albumin therapy will also be documented. The Doppler velocity time integral (VTI) method in estimating stroke volume and cardiac output correlates well with results of concurrent thermodilution cardiac output determinations in patients without significant left-sided valvular regurgitation.
  Cardiac output(CO), Stroke volume (SV), Heart rate (HR)
  CO = [SV * HR]/ 1000
Cardiac output measurement by echocardiography after albumin | Day 2
  Echocardiographic assessment of cardiac output in L/min will be recorded at least 3 time points, day 0, day 1 and day 2.
  The cardiac output at 3 days after enrollment and albumin therapy will also be documented. The Doppler velocity time integral (VTI) method in estimating stroke volume and cardiac output correlates well with results of concurrent thermodilution cardiac output determinations in patients without significant left-sided valvular regurgitation.
  Cardiac output(CO), Stroke volume (SV), Heart rate (HR)
  CO = [SV * HR]/ 1000
Cardiac output measurement by echocardiography after albumin | Day 3
  Echocardiographic assessment of cardiac output in L/min will be recorded at least 3 time points, day 0, day 1 and day 2.
  The cardiac output at 3 days after enrollment and albumin therapy will also be documented. The Doppler velocity time integral (VTI) method in estimating stroke volume and cardiac output correlates well with results of concurrent thermodilution cardiac output determinations in patients without significant left-sided valvular regurgitation.
  Cardiac output(CO), Stroke volume (SV), Heart rate (HR)
  CO = [SV * HR]/ 1000

SECONDARY OUTCOMES:
Change in Cystatin C and Neutrophil gelatinase associated lipocalin (NGAL) level | day 0
Change in NT Pro brain natriuretic peptide (BNP) level | day 0
Change in plasma renin activity level | day 0
Change in Galectin-3 level | day 0
IVC size and collapsibility changes after 20% albumin | Day 0
  IVC maximum and Minimum diameter and collapsibility index determined by percentage change in IVC diameter will be recorded.
IVC size and collapsibility changes after 20% albumin | Day 2
  IVC maximum and Minimum diameter and collapsibility index determined by percentage change in IVC diameter will be recorded.
Lung Ultrasound score change after 20% Albumin | Day 1
IVC size and collapsibility changes after 20% albumin | Day 1
  IVC maximum and Minimum diameter and collapsibility index determined by percentage change in IVC diameter will be recorded.
Lung Ultrasound score change after 20% Albumin | Day 0
Lung Ultrasound score change after 20% Albumin | Day 2

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adebayo D, Neong SF, Wong F. Refractory Ascites in Liver Cirrhosis. Am J Gastroenterol. 2019 Jan;114(1):40-47. doi: 10.1038/s41395-018-0185-6. PMID 29973706
- [Background] Larrue H, Vinel JP, Bureau C. Management of Severe and Refractory Ascites. Clin Liver Dis. 2021 May;25(2):431-440. doi: 10.1016/j.cld.2021.01.010. Epub 2021 Mar 11. PMID 33838859
- [Background] Cardenas A, Arroyo V. Refractory ascites. Dig Dis. 2005;23(1):30-8. doi: 10.1159/000084723. PMID 15920323
- [Background] Salerno F, Guevara M, Bernardi M, Moreau R, Wong F, Angeli P, Garcia-Tsao G, Lee SS. Refractory ascites: pathogenesis, definition and therapy of a severe complication in patients with cirrhosis. Liver Int. 2010 Aug;30(7):937-47. doi: 10.1111/j.1478-3231.2010.02272.x. Epub 2010 May 21. PMID 20492521
- [Result] Izzy M, VanWagner LB, Lin G, Altieri M, Findlay JY, Oh JK, Watt KD, Lee SS; Cirrhotic Cardiomyopathy Consortium. Redefining Cirrhotic Cardiomyopathy for the Modern Era. Hepatology. 2020 Jan;71(1):334-345. doi: 10.1002/hep.30875. Epub 2019 Oct 11. PMID 31342529